CLINICAL TRIAL: NCT04547764
Title: Clinical and Radiographic Evaluation of Triple Antibiotic Paste Pulp Therapy Compared to Vitapex Pulpectomy in Non-vital Primary Molars.
Brief Title: Evaluation of Triple Antibiotic Paste Pulp Therapy Compared to Vitapex in Primary Molars.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Heba sabbagh, assistant professor, King Abdulaziz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 067-16
Record Dates: First submitted 2020-07-11; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Dental Pulp Cavity
Keywords: Deciduous teeth, endodontic treatment, primary molars, pulpectomy.
MeSH Terms: conditions — Dental Caries | interventions — calcium hydroxide, iodoform, silicone oil drug combination; Calcium Hydroxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP group (Experimental)
  Interventions: Drug: triple antibiotic paste (TAP)
- Vitapex group (Active Comparator)
  Interventions: Drug: Vitapex (calcium hydroxide/iodoform paste)

INTERVENTIONS:
Drug: triple antibiotic paste (TAP) — root canal treatment of pulpally involved teeth.
  Arms: TAP group
Drug: Vitapex (calcium hydroxide/iodoform paste) — root canal treatment of pulpally involved teeth.
  Arms: Vitapex group

SUMMARY:
The aim of the study was to compare the clinical and radiographic success of triple antibiotic paste (TAP) which includes (metronidazole, ciprofloxacin, and minocycline) and Vitapex (calcium hydroxide/iodoform paste) for root canal treatment of pulpally involved teeth.

DETAILED DESCRIPTION:
This study evaluated and compared the clinical and radiographic efficacy of non-instrumentation triple antibiotic paste pulp therapy (TAP) versus Vitapex pulpectomy in non-vital primary molars. Healthy 5 to 9 years old children with at least one non-vital primary molar were included in the study. molars were divided based on the subject's cooperation level and parental preference into two groups. In the first group, molars received TAP and in the second group, they received Vitapex pulpectomy followed by a stainless-steel crown. The TAP was freshly prepared and proportioned in equal parts by volume (metronidazole, minocycline, and ciprofloxacin=1:1:1) before the scheduled treatment appointment. The clinical and radiographic examination was performed by two calibrated and trained pediatric dentists at the pre-operative baseline and at the six- and 12-months follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Primary molars with at least one of the following signs and symptoms were eligible and were included in the study:

* badly decayed with signs of irreversible pulpitis,
* necrosis and chronic infection such as: pain or tenderness to percussion and palpation, abscess, fistula-opening, gingival swelling, grade II and greater pathological tooth mobility, evidence of periapical/bifurcation radiolucency,

All the teeth included, had physiological root resorption of less than one third of the root.

Exclusion Criteria

* Teeth showing radiographic evidence of excessive internal or external root resorption,
* perforated pulpal floor,
* excessive bone loss in furcation area involving the underlying tooth germ,
* non- restorable teeth were excluded from the study.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
fissure-exact test | up to 12 months
  The success rate of case and control groups, at 6 and 12 months follow-ups, are compared by Fissure-Exact Test.

CONTACTS AND LOCATIONS:
Overall Officials: heba sabbagh, PhD, Principal Investigator — Assistant Professor, Department of Pediatric Dentistry King Abdulaziz University
Locations (1):
- King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia